CLINICAL TRIAL: NCT00004251
Title: A Phase II Study of Letrozole in Patients With Advanced or Recurrent Endometrial Cancer
Brief Title: Letrozole in Treating Women With Recurrent or Metastatic Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I126; CAN-NCIC-IND126 (Other: PDQ); NOVARTIS-FEM-CA-02 (Other: Novartis); CDR0000067498 (Other: PDQ)
Record Dates: First submitted 2000-01-28; First posted 2004-06-17 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Endometrial Cancer
Keywords: stage IV endometrial carcinoma; recurrent endometrial carcinoma; endometrial adenocarcinoma; endometrial adenosquamous cell carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Letrozole (Experimental): Letrozole 2.5 mg po daily
  Interventions: Drug: letrozole

INTERVENTIONS:
Drug: letrozole — 2.5 mg of letrozole per day

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of letrozole in treating women who have recurrent or metastatic endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of letrozole, in terms of objective tumor response and time to progression, in women with recurrent or metastatic endometrial cancer. II. Determine the toxicity of letrozole in these patients. III. Determine the relationship between tumor receptor status, histologic grade, tumor aromatase activity, and tumor response in these patients.

OUTLINE: Patients receive an oral letrozole tablet daily. Treatment continues for patients with complete or partial response until disease progression or unacceptable toxicity. Patients with stable disease may discontinue therapy after 24 weeks. Patients are followed at 1 month and then every 3 months until death.

PROJECTED ACCRUAL: Up to 30 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven, recurrent or metastatic, adenocarcinoma or adenosquamous carcinoma of the endometrium not curable by surgery and/or radiotherapy Failed one prior progestin therapy for advanced/metastatic disease OR Considered for letrozole as first line therapy of advanced/metastatic disease No clear cell or papillary serous histology, uterine sarcomas, mixed muellerian tumors, and/or adenosarcomas At least one site of measurable disease by clinical exam, CT, or MRI scan Bone lesion(s) are not considered measurable No CNS metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Menopausal status: Postmenopausal (surgical or natural) Life expectancy: At least 12 weeks Hematopoietic: Absolute granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than upper limit of normal (ULN) AST or ALT no greater than 2 times ULN Alkaline phosphatase less than 2 times ULN Renal: Creatinine no greater than 2 times ULN Other: No other malignancy within the past 5 years, except: Adequately treated basal or squamous cell skin cancer Carcinoma in situ of the cervix No other concurrent medical illness that would preclude compliance

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for advanced/metastatic disease At least 4 weeks since prior adjuvant chemotherapy Endocrine therapy: See Disease Characteristics No more than one prior progestational hormone therapy regimen for advanced/metastatic disease At least 1 week since prior hormonal therapy No prior tamoxifen or other aromatase inhibitor therapy Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiotherapy Concurrent radiotherapy for symptomatic metastatic lesions allowed Surgery: See Disease Characteristics Other: No other concurrent anticancer therapy No other concurrent investigational therapy

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2000-01-19 (Actual); Primary Completion 2002-09-13 (Actual); Study Completion 2011-01-18 (Actual)

PRIMARY OUTCOMES:
Objective tumour response | 3 years

SECONDARY OUTCOMES:
duration of response and time to progression | 3 years
toxicity | 3 years
tumour response | 3 years
  Correlation of tumour response with pre-treatment ER/PR status, histological grade and aromatase levels.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Fyles, MD, Study Chair — Princess Margaret Hospital, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ma BB, Oza A, Eisenhauer E, Stanimir G, Carey M, Chapman W, Latta E, Sidhu K, Powers J, Walsh W, Fyles A. The activity of letrozole in patients with advanced or recurrent endometrial cancer and correlation with biological markers--a study of the National Cancer Institute of Canada Clinical Trials Group. Int J Gynecol Cancer. 2004 Jul-Aug;14(4):650-8. doi: 10.1111/j.1048-891X.2004.14419.x. PMID 15304161
- [Result] Sidhu K, Fyles A, Eisenhauer E, et al.: Phase II study of the aromatase inhibitor letrozole in endometrial carcinoma - NCIC CTG IND 126. [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-2520, 2001.